CLINICAL TRIAL: NCT04301921
Title: Strategies to Maintain Radial Artery Patency Following Diagnostic Coronary Angiography - Diagnostic Transradial Coronary Angiography Without Systemic Anticoagulatio
Acronym: RAPID-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Senior physician, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAPID-1
Record Dates: First submitted 2020-02-18; First posted 2020-03-10 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Patients Undergoing Diagnostic Coronary Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Traditional puncture site + no anticoagulation
  Interventions: Other: Traditional punkcture site and No anticoagulation
- Group 2 (Other): Traditional puncture site + ACT-guided anticoagulation
  Interventions: Other: Traditional punkcture site and ACT-guided anticoagulation

INTERVENTIONS:
Other: Traditional punkcture site and No anticoagulation — Traditional punkcture site and No anticoagulation
  Arms: Group 1
Other: Traditional punkcture site and ACT-guided anticoagulation — Traditional punkcture site and ACT-guided anticoagulation
  Arms: Group 2

SUMMARY:
To investigate whether omitting systemic anticoagulation during transradial coronary angiography and/or a distal radial access reduce the risk of postprocedural radial artery occlusion

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication to perform diagnostic coronary angiography
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Preexisting or already administered anticoagulation prior to coronary angiography
* Planned coronary intervention
* Preexisting radial artery occlusion or missing pulse at the potential puncture sites
* Allergy / intolerance to anticoagulants
* Active bleeding or comorbidity with elevated bleeding risk
* Pregnancy
* Inability to sign informed consent
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postprocedural RAO | Day 1
  Will be the occurrence of postprocedural RAO assessed with high-resolution vascular ultrasound. Experienced sonographers will perform color Doppler ultrasound in all study patients after removal of the compression device to examine the radial, ulnar, and brachial arteries of the access forearm.
Bleeding events | Day 1
  Will be bleeding events according to Bleeding Academic Research Consortium (BARC) criteria.

SECONDARY OUTCOMES:
Sonographic characteristics of radial artery occlusion | 3 Month
  Occlusion lengths or minimal residual perfusion

REFERENCES:
- [Derived] Stiermaier T, Grunewalder M, Patz T, Rawish E, Joost A, Meusel M, Marquetand C, Kurz T, Schmidt T, Frerker C, Fuernau G, Eitel I. Distal access and procedural anticoagulation to prevent radial artery occlusion after coronary angiography - the randomised RAPID trial. EuroIntervention. 2025 Apr 7;21(7):e366-e375. doi: 10.4244/EIJ-D-24-00846. PMID 40191883